CLINICAL TRIAL: NCT05402930
Title: Usefulness of Angiomammography for Predicting the Response to Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: Angiomammography and Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-4433
Record Dates: First submitted 2022-05-20; First posted 2022-06-02 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy (Experimental)
  Interventions: Diagnostic Test: Angiomammography

INTERVENTIONS:
Diagnostic Test: Angiomammography — Patients will receive their care in a standard manner. Breast MRI is one modality used by physicians to monitor response to neoadjuvant chemotherapy and will therefore be used as standard. A CESM exam will be added at the same time as the MRI.
  Patients will have a physical exam, breast MRI and CESM before the start of chemotherapy (less than 2 weeks). These examinations will be repeated after cycle 2 (±1 week) and at the end of chemotherapy. After each cycle of chemotherapy, the tumor will be measured in two axes by the attending physician.
  Histological examination of the surgical specimen will be used to determine the pCR. Responses observed on MRI and CESM will be compared to pCR.

SUMMARY:
The best prognostic factor following neoadjuvant chemotherapy is the pathological complete response (pCR). pCR is defined as the absence of invading cells in the breast and lymph nodes following neoadjuvant chemotherapy treatment. Since patients with pCR have a better prognosis than those without pCR, some studies have evaluated different methods to predict pCR early in treatment. Thus, patients who do not respond optimally to treatment could be identified early and changed treatment in order to maximize the chances of pCR and avoid the morbidity of poorly effective treatments. To do this, several modalities have been proposed, including MRI, mammography, ultrasound, positron emission tomography, elastography, and serial biopsies, but these techniques have shown predictive and sometimes expensive. Nevertheless, assessment of tumor response after cycle 2 has been suggested to be appropriate for the prediction of pCR.

The main objective of this study is to compare the performance of two diagnostic modalities, namely CESM and MRI, in the evaluation of the response of a malignant breast tumor to neoadjuvant chemotherapy and the prediction of pCR. The radiological response will also be compared to the clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 and over
* Histologically proven breast cancer by large gauge needle
* No evidence of distant metastasis
* Neoadjuvant chemotherapy with or without concomitant targeted therapy
* Breast tumor initially measurable by clinical examination

Exclusion Criteria:

* Refusal to perform the biopsy or surgery
* Pregnant or possibly pregnant woman
* Usual contraindication to contrast product

  * Significant kidney failure
  * Allergy to contrast medium
* frank hyperthyroidism
* Usual contraindications to MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a pCR accoreding to angiomammography, based on a 50% reduction in lesion size at angiomammography | Cycle 2 (each cycle being 21 days), i.e., after the chemotherapy on day 1 of cycle 2 and before cycle 3.
  Prediction of pCR using angiomammography after cycle 2 of neoadjuvant chemotherapy, based on a 50% reduction in lesion size at angiomammography

CONTACTS AND LOCATIONS:
Locations (1):
- St-Sacrement Hospital, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No